CLINICAL TRIAL: NCT00617864
Title: The Effect of Human Albumin Infusion on VEGF Levels in Women at Risk for Ovarian Hyperstimulation Syndrome.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The syndrome of hyperstimulation is so rare that after one year no patients were eligible.The study was withdrawn and never started.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0707002880
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Ovarian Hyperstimulation Syndrome
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group will receive infusion of human albumin
  Interventions: Drug: Human Albumin Infusion
- 2 (Placebo Comparator): Group will receive infusion of saline
  Interventions: Drug: Saline Infusion

INTERVENTIONS:
Drug: Human Albumin Infusion — Group will receive single infusion of albumin at the time of oocyte retrieval.
  Arms: 1
Drug: Saline Infusion — Group will receive single infusion of saline at the time of oocyte retrieval.
  Arms: 2

SUMMARY:
This research study was designed to look at the effect of human albumin transfusion on circulating levels of Vascular Endothelial Derived Growth Factor (VEGF), a protein that is believed to be responsible for the syndrome of ovarian hyperstimulation. Patients have been asked to participate because they are identified as at risk for the Ovarian Hyperstimulation Syndrome (OHSS), a potentially serious complication of in vitro fertilization. It has been established that the onset of OHSS may be preventable by the infusion of albumin at the time of egg retrieval; however, we do not know by what mechanism albumin works. As we know the pathogenesis of OHSS is related to VEGF released from the ovaries, we believe human albumin may serve to "bind up" this VEGF and prevent it from causing its harmful effects. The purpose of this study is to evaluate the effect of albumin infusion on blood and urine VEGF levels in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients undergoing in vitro fertilization with or without ICSI
* Estradiol > 3000 pg/mL at the time of hCG administration
* >/= 20 follicles seen during ultrasound monitoring
* Patients with polycystic ovarian syndrome

Exclusion Criteria:

* Patients with only one ovary
* Patients with medical contraindication to human albumin (hypersensitivity, hypervolemia, cardiac insufficiency, hypertension, esophageal varices, pulmonary edema, severe anemia, renal failure)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09

PRIMARY OUTCOMES:
Serum VEGF levels | Time surrounding egg retrieval

SECONDARY OUTCOMES:
Urine VEGF levels | Time surrounding egg retrieval
Pregnancy | Time surrounding egg retrieval

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Patrizio, MD, MBE, HCLD, Principal Investigator — Yale University
Locations (1):
- Yale Fertility Center, New Haven, Connecticut, United States